CLINICAL TRIAL: NCT00537537
Title: An Open Label, Response Adaptive Study of Telbivudine in Adults With HBeAg Positive Compensated CHB
Brief Title: To Evaluate Antiviral Efficacy of Telbivudine in Hepatitis B Antigen Positive (HbeAg-positive) Compensated Chronic Hepatitis B (CHB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600AIN01
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2016-04

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic, Hepatitis B e Antigen positive, Adults, Telbivudine, Adefovir
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Bronchiolitis Obliterans Syndrome | interventions — Telbivudine

ARMS (3):
- 1 (Active Comparator): Telbivudine
  Interventions: Drug: Telbivudine
- 2 (Active Comparator): Telbivudine
  Interventions: Drug: Telbivudine
- 3 (Active Comparator): Telbivudine
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Telbivudine

SUMMARY:
This study is to evaluate the antiviral efficacy of add-on adefovir to telbivudine in non-responders to telbivudine monotherapy after 24 and 36 initial weeks. Antiviral efficacy is assessed by hepatitis B virus (HBV) DNA non-detectability (PCR <300 copies/ml) by week 104 with CHB.

ELIGIBILITY:
Inclusion Criteria:

Male or female, at least 18 yrs of age; HBsAg positive, HBeAg positive and anti-HBe negative at the time of screening; Quantifiable serum HBV DNA levels of >105copies/ml; ALT levels any level; Treatment naïve; Baseline liver histology in case of ALT levels within normal limits performed within last 12 months) indicative of chronic hepatitis B changes Metavir score F >2; Willing and able to comply with the study drug regimen and all other study requirements; The patient or guardian is willing and able to explore written informed consent to participate in the study. Exclusion Criteria:

Patient is pregnant or breastfeeding. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (HCG) at Screening visit; Patient is of childbearing potential (men and women) and unwilling to use a barrier method of contraception. It is required that a barrier method of contraception be used (i.e. condom with spermicide or diaphragm with spermicide) by patients of childbearing potential (men and women) regardless of whether a hormonal agent also is used as a method of contraception; Patient is co infected with hepatitis C virus (HCV), HIV. Patients will be tested for antibodies to HCV & HIV in the Screening assessments;Patient has a medical condition that requires prolonged or frequent use of systemic acyclovir or famciclovir; Patient is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years; Patient has a medical condition that requires frequent or prolonged use of systemic corticosteroids; Patients who has been on warfarin or other anticoagulants during 30 days prior to screening or if expected during the present study; Patient has any other concurrent medical condition, at clinician's discretion, likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Antiviral efficacy with adefovir combination assessed by HBV DNA non-detectability (PCR <300 copies/ml) by week 104.

SECONDARY OUTCOMES:
Antiviral efficacy with telbivudine alone assessed by HBV DNA non-detectability (PCR <300 copies/ml) at week 24 and 36.
HBeAg loss & HBeAg seroconversion (defined as a loss of HBeAg and a gain of detectable level of HBeAb).
Alanine Transaminase (ALT) normalization, in patients with raised levels at baseline.
Change in HBV DNA level (log10 copies/ml) from baseline to week 4, 8, 12, 24, 36, 52, 76 and 104.
Viral breakthrough, defined as increase of HBV DNA by 1 log10 copies/ml from treatment nadir, at any point after week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (3):
- India (3):
  - Novartis Investigative Site, Hyderabad
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, Vellore